CLINICAL TRIAL: NCT02393677
Title: Supraclavicular Brachial Plexus Block Using Ropivacaine Alone or Combined With Dexmedetomidine for Upper Limb Surgery: A Prospective, Randomized, Double-blinded, Comparative Study
Brief Title: Supraclavicular Brachial Plexus Block Using Ropivacaine Alone and With Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Bikramjit Das, Assistant Professor, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DN57/FM
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Brachial Plexus Anesthesia
MeSH Terms: interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Placebo Comparator): amide local anesthetic
  Interventions: Drug: Ropivacaine
- Ropivacaine with Dexmedetomidine (Active Comparator): combination of amide local anaesthetic and alpha2 agonist
  Interventions: Drug: Ropivacaine with Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine 0.5% 30 ml was used to block brachial plexus
  Other Names: Ropin
  Arms: Ropivacaine
Drug: Ropivacaine with Dexmedetomidine — Dexmedetomidine 1 microgram per kilogram bodyweight was added with 30 ml 0.5% Ropivacaine to block brachial plexus
  Other Names: Ropin with Dextomid
  Arms: Ropivacaine with Dexmedetomidine

SUMMARY:
80 American Society of Anesthesiologists (ASA) grade I-II patients, 18-60 years old,scheduled for elective upper limb orthopaedic surgery under supraclavicular brachial plexus block, were included in this prospective study. The patients were randomly assigned to group R (Ropivacaine alone) and group RD (Ropivacaine and dexmedetomidine) (40 patients in each group). Group R received Ropivacaine 0.50% (30 cc) + placebo and group RD received Ropivacaine 0.50% (30 cc) + dexmedetomidine 1 µg/kg.

DETAILED DESCRIPTION:
After Institutional Ethical Committee approval and written informed consent, a prospective, randomized, double-blinded study was carried out on 80 ASA Grade I and II patients of either sex, aged 18-60 years, undergoing various orthopaedic surgeries on the upper limb under supraclavicular brachial plexus block. A power analysis was performed to determine the necessary number of patients for each group based on duration of analgesia. With a 2-sided type I error of 5% and study power at 80%, it was estimated that 38 patients would be needed in each group in order to detect a difference of 35 min in the duration of analgesia between the 2 groups. The study was conducted in two groups of 40 patients each. Patients were randomly chosen by computer-generated random selection to one of the following groups:

Group R: Ropivacaine 0.50% (30 cc) + Placebo Group RD: Ropivacaine 0.50% (30 cc) + Dexmedetomidine 1 µg/kg Randomization was performed by an independent statistician and concealed from patients and investigators until completion of statistical analysis. Patients were instructed preoperatively about use of the verbal rating scale (VRS) for pain assessment (VRS: 0 = no pain, 10=worst pain possible). On arrival in the operation room, baseline heart rate, blood pressure and oxygen saturation were recorded. An intravenous line was secured in the unaffected limb and Ringer's lactate was started. Patients were given midazolam intravenous (IV) (0.03 mg/kg) as premedication 10-15 min before beginning each blocks technique. Subcutaneous injection with 2 mL of 2% lidocaine was administered at the needle insertion site. All the patients received brachial plexus block through the supraclavicular approach by an experienced anesthesiologist different from the one assessing the patient intra- and post-operatively. Both were blinded to the treatment groups. Neural localization was achieved by using a nerve locator (Stimuplex® Dig RC, B.Braun, Melsungen AG, Melsungen, Germany) connected to a 22 G, 50-mm-long stimulating needle (Stimuplex, Braun, Germany). The location end point was a distal motor response with an output lower than 0.5 milliampere (mA).

Following negative aspiration, 30 mL of a solution containing local anesthetic combined with placebo or dexmedetomidine as mentioned above was injected and the use of Dexmedetomidine was off-label. A 5-min compression was performed to facilitate an even drug distribution. Sensory blockade was assessed every 3 min and motor block was evaluated every 5 min within the first 30 min following completion of drug administration. Sensory block was confirmed by pinprick sensation using a 23-G needle in all dermatomes of the brachial plexus (C5-T1) i.e. median nerve, radial nerve, ulnar nerve and musculocutaneous nerve. Sensory onset was considered when there was a dull sensation to pin prick along the distribution of any of these nerves (Grade 1). Complete sensory block was considered when there was complete loss of sensation to pin prick.

Sensory block was graded as- Grade 0 Sharp pin felt Grade 1 Analgesia, dull sensation felt Grade 2 Anesthesia, no sensation felt

Motor blockade was evaluated by the ability to flex the elbow and hand against gravity as follows :

Grade 1 Ability to flex and extend the forearm Grade 2 Ability to flex or extend only the wrist and fingers Grade 3 Ability to flex or extend only the fingers Grade 4 Inability to move the forearm, wrist, and fingers Onset of motor block was defined as the time from injection of local anesthetic mixture until achieving a reduction in motor power to grade 3 or less. The block was considered incomplete when any of the segments supplied by median, radial, ulnar and musculocutaneous nerve did not have analgesia even after 30 min of drug injection. These patients were supplemented with intravenous fentanyl (2 μg/ kg) and midazolam (0.03 mg/kg). When more than one nerve remained unaffected, it was considered a failed block. In this case, general anesthesia was given intraoperatively. Patients were monitored for hemodynamic variables such as heart rate, blood pressure and oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* 80 ASA Grade I and II patients of either sex, aged 18-60 years, undergoing various orthopaedic surgeries on the upper limb under supraclavicular brachial plexus block.

Exclusion Criteria:

* Patient refusal
* Patients with chronic pain (pain lasting more than 12 weeks)
* Those using chronic analgesic medications (opioid, non steroidal anti-inflammatory drugs, anticonvulsants, antidepressants)
* Coagulopathy
* History of brachial plexus injury
* Allergy to the study drugs
* Patients taking other medications with α-adrenergic blocking effect
* Hepatic or renal insufficiency
* Systemic infection or infection at the site of injection, and shoulder surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahin N Jamil, MD, Study Director — Professor, Aligarh Muslim University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine | Ropivacaine With Dexmedetomidine
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine | Ropivacaine With Dexmedetomidine | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (9.6) | 34.52 (12.8) | 34.86 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 20 | 17 | 37
Region of Enrollment [Number; unit: participants]
  India | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia
Time Frame: upto 8 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ropivacaine | Ropivacaine With Dexmedetomidine
Number analyzed (Participants) | 40 | 40
minutes | 413.73 (89.92) | 197.35 (28.67)

2. Secondary Outcome: Onset of Sensory Block
Time Frame: 20 minutes
Reporting Status: Not Posted

3. Secondary Outcome: Onset of Motor Block
Time Frame: 30minutes
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Motor Block
Time Frame: 6 hours
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Haemodynamic Changes
Time Frame: 8 hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Complications
Time Frame: 2 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ropivacaine | Ropivacaine With Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 4/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine (N=40) | Ropivacaine With Dexmedetomidine (N=40)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes